CLINICAL TRIAL: NCT00817115
Title: Trial to Determine Non-inferiority of Exposure Dose Reduction and Diagnostic Performance of Region-of-Interest Fluoroscopy (X-ray Fovea Imaging) Compared to Standard Fluoroscopy in Patients Undergoing Cardiac Interventional Procedures
Brief Title: Evaluation of Exposure Reduction Using Region-of-Interest Fluoroscopy (X-ray Fovea Imaging) in Cardiac Interventions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: General Electric (Industry)
Responsible Party: Dr. Alexander Dick, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 005-2008
Record Dates: First submitted 2008-11-14; First posted 2009-01-06 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-01

CONDITIONS: Cardiovascular Diseases
Keywords: Region-of-Interest Imaging; X-ray Fovea Imaging; Cardiovascular Diseases; Radiation Dosage; Radiographic Image Enhancement; Radiography, Interventional
MeSH Terms: conditions — Cardiovascular Diseases

ARMS (2):
- 1 (No Intervention): Subjects undergoing routine cardiac catheterization or interventional procedures using the standard fluoroscopy system.
- 2 (Experimental): Subjects undergoing routine cardiac catheterization or interventional procedures using the region-of-interest fluoroscopy (x-ray fovea imaging) system.
  Interventions: Device: Region-of-Interest Imaging (X-ray Fovea Imaging)

INTERVENTIONS:
Device: Region-of-Interest Imaging (X-ray Fovea Imaging) — Use of an experimental fluoroscopy system fitted with a region-of-interest attenuator (fovea) to evaluate or treat lesions during cardiac interventional procedures.
  Arms: 2

SUMMARY:
The aim of the proposed study is to compare the exposure dose and diagnostic performance of region-of-interest fluoroscopy compared to standard fluoroscopy in patients and interventionists during cardiac interventional procedures. It is hypothesized that systematic application of x-ray attenuation will significantly reduce the radiation exposure of the interventional procedure while maintaining image quality, thereby decreasing risk to the patient.

DETAILED DESCRIPTION:
X-ray catheterization is used to guide minimally invasive procedures including percutaneous coronary interventions (PCIs), involving diffuse and multiple vessel disease and total chronic occlusion as well as electrophysiology (EP) procedures. While the medical benefit to patients outweighs the procedural risk, long fluoroscopy times associated with complex interventions have resulted in acute radiation injuries to patients. Radiation induced cancers have also become a concern in younger patient populations. With the increased number, diversity and complexity of the interventions performed, there has been a growing interest in reducing the long-term exposure risk to medical personnel (interventionists).

Conventional methods to reduce in radiation exposure, however, impact and often degrade diagnostic image quality. Catheterization procedures focus on a small portion of the anatomy forming the central region of the image with the periphery providing contextual information. Thus, decreasing the image quality in periphery can provide an overall exposure reduction to patients and interventionists without impacting on diagnosis. This can be achieved by introducing a pre-patient region-of-interest (ROI) attenuator that collimates the primary x-ray beam, reducing exposure to peripheral regions and decreasing integral radiation to the patient and scatter radiation to the interventionist.

The goal of this study is to investigate the exposure dose reduction provided by ROI imaging to patients and interventionists undergoing catheterization and to examine the feasibility of using the ROI attenuator in routine clinical practice for future integration into commercial x-ray imaging systems. The aim is to obtain exposure dose data and cardiac angiography images from subjects undergoing routine interventional procedures performed with and without ROI attenuation (experimental and control groups, respectively). For the experimental group, the interventionists performing the procedure will determine the appropriate application of the ROI attenuator and the duration of its use on specific patient lesions. An internal pilot study will be initially conducted on approximately 30 patients (15 per group) to obtain estimates on patient and operator dose reduction and variability. The on-going clinical trial will then be performed on an additional 40 patients (where the final protocol procedures and recruitment will be refined based on results from the pilot study).

ELIGIBILITY:
Inclusion Criteria:

* The subject is greater than 18 years of age.
* The subject is currently planned for conventional cardiac interventional procedures (i.e. catheterization, percutaneous coronary intervention (PCI), electrophysiology (EP) ablations and procedures) as specified by his/her physician.
* The subject is able and willing to comply with study procedures, and signed and dated informed consent is obtained.

Exclusion Criteria:

* The subject is pregnant or trying to become pregnant.
* The subject requires urgent/emergent cardiac catheterization, PCI, and/or EP procedures as per treating physician.
* The subject has been previously included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
X-ray exposure area product, primary and scatter radiation to patient and interventionist and procedure and irradiation time for interventions performed without and with region-of-interest imaging (control and experimental arms, respectively). | The outcome measure will be recorded per patient procedure. A comparison between control and experimental arms will be conducted after the pilot study (at ~1 to 2 months) and at end the full study (at ~4 to 6 months).

SECONDARY OUTCOMES:
Quality and diagnostic benefit of images obtained without and with the region-of-interest imaging. | Retrospective expert comparison of images from patient procedures (between control and experimental arms) will occur within 1 to 3 months after the completion of the pilot study and the full study.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander J Dick, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Normand Robert, PhD, Study Director — Sunnybrook Health Sciences Centre; John A Rowlands, PhD, Study Chair — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada